CLINICAL TRIAL: NCT03180749
Title: Post-Marketing Clinical Follow-up of an Anular Closure System (Barricaid®) to Confirm Comparability of Outcome Between Devices With Subcomponents From Two Different Suppliers
Brief Title: Post-Marketing Clinical Follow-Up of a Spine Implant
Acronym: PMCFU
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Intrinsic Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: EUBARD-CP-001-PMCFU
Record Dates: First submitted 2017-06-06; First posted 2017-06-08 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Lumbar Disc Herniation; Annular Tear of Lumbar Disc
MeSH Terms: conditions — Intervertebral Disc Displacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients implanted with vendor B anchor
  Interventions: Other: Follow up per standard of care

INTERVENTIONS:
Other: Follow up per standard of care — Patients will come in 2 years post implantation and receive standard examinations

SUMMARY:
Post-Marketing Clinical Follow-up of an Anular Closure System (Barricaid®) to Confirm Comparability of Outcome between Devices with Subcomponents from Two Different Suppliers

DETAILED DESCRIPTION:
Comparison of device integrity (anchor fracture and/or mesh detachment) and device movement/migration in patients implanted with the Barricaids with anchors from two different suppliers.

ELIGIBILITY:
Inclusion Criteria:

* Each site will enroll all patients who were implanted with a Barricaid with an anchor manufactured by the second manufacturer.
* Patients must be 18 years of age or older and able to understand and consent to participate in the study.

Exclusion Criteria:

* Not defined

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Sites will enroll all eligible patients who were implanted with the Barricaid with an anchor of the second vendor (identifiable via the lot number), and consent to participate.
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2017-03-02 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Device failures | 22+ months post implantation
  Device failures and movement/migration will be assessed by a radiographic core laboratory.

CONTACTS AND LOCATIONS:
Locations (6):
- Germany (5):
  - Wirbelsäulenzentrum Bielefeld, Bielefeld
  - Klinikum Itzehoe, Itzehoe
  - Universitaetsklinikum Schleswig-Holstein, Kiel
  - Bonifatius Hospital Lingen, Lingen
  - UKM Marienhospital Steinfurt, Steinfurt
- Orthopädie St.Gallen, Sankt Gallen, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided